CLINICAL TRIAL: NCT07232602
Title: A Phase 1/2 Open-Label Rolling-Arm Umbrella Platform Study of Investigational Agents in Combination With Enfortumab Vedotin Plus Pembrolizumab as First-Line Treatment in Participants With Locally Advanced or Metastatic Urothelial Carcinoma: KEYMAKER-U04-Substudy 04D
Brief Title: KEYMAKER-U04 Substudy 04D: A Clinical Study of New Treatments Given With Enfortumab Vedotin and Pembrolizumab in People With Urothelial Cancer (MK-3475-04D/KEYMAKER-U04)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-04D; U1111-1322-3713 (Registry Identifier: UTN); 2025-522253-19-00 (Registry Identifier: EU CT); MK-3475-04D (Other: MSD)
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — enfortumab vedotin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm A: MK-3120 + Enfortumab Vedotin (EV) + Pembrolizumab (Experimental): Participants will receive MK-3120 administered intravenously on Day 1 and Day 8 of each 3-week cycle and EV administered intravenously on Day 1 and Day 8 of each 3-week cycle until documented disease progression or any other discontinuation criterion is met and Pembrolizumab 200 mg administered intravenously on Day 1 of each 3-week cycle for up to 35 cycles (~2 years).
  Interventions: Drug: MK-3120; Drug: EV; Biological: Pembrolizumab; Drug: Rescue Medication

INTERVENTIONS:
Drug: MK-3120 — Administered via intravenous (IV) infusion on day 1 and day 8 of each 3-week cycle
Drug: EV — Administered via IV infusion on day 1 and day 8 of each 3-week cycle
  Other Names: AGS 22M6E; AGS-22CE
Biological: Pembrolizumab — Administered via IV infusion on day 1 of each 3-week cycle
  Other Names: MK-3475; KEYTRUDA®
Drug: Rescue Medication — Participants receive rescue medication at the investigator's discretion, per approved product label. Recommended rescue medication is Granulocyte Colony-Stimulating Factor (G-CSF).

SUMMARY:
Researchers are looking for new ways to treat people with urothelial cancer (UC) that is locally advanced or metastatic. The standard treatment for locally advanced or metastatic UC is enfortumab vedotin (EV) given with pembrolizumab.

The goals of this study are to learn about:

* The safety of the study treatment when given with standard treatment and if people tolerate it
* The number of people who have the cancer respond (cancer gets smaller or goes away) with the new study treatment when given with standard treatment.

DETAILED DESCRIPTION:
This is a substudy of the master protocol MK-3475-U04 (KEYMAKER-U04)

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has histologically documented urothelial carcinoma (UC) that is locally advanced and unresectable or metastatic
* Must provide a newly obtained or archival tumor tissue sample (core or excisional biopsy)
* Must not have received prior systemic therapy for locally advanced or metastatic UC
* If infected with Human Immunodeficiency Virus (HIV), has well controlled HIV on antiretroviral therapy
* If positive for hepatitis B surface antigen, has received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and has undetectable HBV viral load before randomization
* If participant has a history of hepatitis C virus (HCV), has undetectable HCV viral load before randomization

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has history of documented severe dry eye syndrome, severe Meibomian gland disease and/or blepharitis, or corneal disease that prevents/delays corneal healing
* Has active keratitis or corneal ulcerations
* Has active inflammatory bowel disease requiring immunosuppressive medication, or previous history of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis, or chronic diarrhea)
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease within the 6 months preceding study intervention
* Has a history of uncontrolled diabetes
* Has pleural effusion, ascites, and/or pericardial effusion that are symptomatic or require repeated drainage
* Has active autoimmune disease that has required systemic treatment in the past 2 years
* Has known additional malignancy that is progressing or has required active treatment within the past 2 years
* Has known active central nervous system metastases and/or carcinomatous meningitis
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids, or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy
* If infected with HIV, has a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has concurrent active HBV and HCV infection
* Has a history of stem cell/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2030-10-18 (Estimated); Study Completion 2030-10-18 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 27 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants that experience AEs will be reported.
Number of Participants Who Experience a Dose Limiting Toxicity (DLT) | Up to approximately 21 days
  DLT will be defined as any drug-related AE observed during the DLT evaluation period that results in a change to a given dose or a delay in initiating the next treatment. The number of participants who experience a DLT as Assessed Using Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 will be presented.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 24 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants that discontinue study intervention due to an AE will be reported.
Objective Response Rate (ORR) as Assessed by Investigator | Up to approximately 58 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experience CR or PR as assessed by Investigator will be presented.

SECONDARY OUTCOMES:
Duration of Response (DOR) as Assessed by Investigator | Up to approximately 58 months
  For participants who demonstrate a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1), DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by investigator will be presented.
Serum Maximum Concentration (Cmax) of MK-3120 Antibody-Drug Conjugate (ADC) | Predose and at designated time points post-dose (up to approximately 24 months)
  Cmax is defined as the peak concentration over the dosing interval. Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine Cmax of MK-3120 ADC.
Serum Trough Concentration (Ctrough) of MK-3120 ADC | Predose and at designated time points post-dose (up to approximately 24 months)
  Ctrough is defined as the trough concentration. Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine Ctrough of MK-3120 ADC.
Serum Cmax of MK-3120 Total Antibodies (TAb) | Predose and at designated time points post-dose (up to approximately 24 months)
  Cmax is defined as the peak concentration over the dosing interval. Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine Cmax of MK-3120 TAb.
Serum Ctrough of MK-3120 TAb | Predose and at designated time points post-dose (up to approximately 24 months)
  Ctrough is defined as the trough concentration. Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine Ctrough of MK-3120 TAb.
Plasma Cmax of MK-3120 Free Payload | Predose and at designated time points post-dose (up to approximately 24 months)
  Cmax is defined as the peak concentration over the dosing interval. Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine Cmax of MK-3120 Free Payload.
Plasma Ctrough of MK-3120 Free Payload | Predose and at designated time points post-dose (up to approximately 24 months)
  Ctrough is defined as the trough concentration. Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine Ctrough of MK-3120 Free Payload.
Serum Cmax of EV ADC | Predose and at designated time points post-dose (up to approximately 24 months)
  Cmax is defined as the peak concentration over the dosing interval. Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine Cmax of EV ADC.
Serum Ctrough of EV ADC | Predose and at designated time points post-dose (up to approximately 24 months)
  Ctrough is defined as the trough concentration. Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine Ctrough of EV ADC.
Serum Cmax of EV TAb | Predose and at designated time points post-dose (up to approximately 24 months)
  Cmax is defined as the peak concentration over the dosing interval. Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine Cmax of Enfortumab Vedotin (EV) TAb.
Serum Ctrough of EV TAb | Predose and at designated time points post-dose (up to approximately 24 months)
  Ctrough is defined as the trough concentration. Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine Ctrough of EV TAb.
Plasma Cmax of EV Free Payload | Predose and at designated time points post-dose (up to approximately 24 months)
  Cmax is defined as the peak concentration over the dosing interval. Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine Cmax of Enfortumab Vedotin (EV) Free Payload.
Plasma Ctrough of EV Free Payload | Predose and at designated time points post-dose (up to approximately 24 months)
  Ctrough is defined as the trough concentration. Blood samples collected pre-dose and at multiple timepoints post-dose will be used to determine Ctrough of EV Free Payload.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- Israel (2):
  - Rambam Health Care Campus ( Site 5501), Haifa
  - Rabin Medical Center ( Site 5504), Petah Tikva

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/